CLINICAL TRIAL: NCT03696992
Title: Blue Laser Imaging Versus Narrow Band Imaging Versus White Light Imaging for Detection of Adenoma in the Proximal Colon: A Prospective Randomized Study
Brief Title: BLI, NBI or White Light Colonoscopy for Proximal Colonic Adenoma
Acronym: BNW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, LEUNG Wai Keung, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: UW18-420
Record Dates: First submitted 2018-09-27; First posted 2018-10-05 (Actual); Last update posted 2022-04-21 (Actual); Status verified 2022-04

CONDITIONS: Colon Adenoma
Keywords: colonoscopy

STUDY DESIGN:
Intervention Model Description: Prospective randomized design
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NBI (Experimental): Tandem colonoscopy with NBI follow by WL
  Interventions: Procedure: Tandem colonoscopy
- BLI (Active Comparator): Tandem colonoscopy with BLI follow by WLI
  Interventions: Procedure: Tandem colonoscopy
- WLI (Experimental): Tandem colonoscopy with WLI follow by WL
  Interventions: Procedure: Tandem colonoscopy

INTERVENTIONS:
Procedure: Tandem colonoscopy — Tandem colonoscopy with different image modalities

SUMMARY:
This is a prospective randomised trial comparing the proximal adenoma detection rate and miss rate by blue laser imaging (BLI), narrow band imaging or white light colonoscopy.

DETAILED DESCRIPTION:
Study population:

Consecutive adult patients, age 40 or above, undergoing outpatient colonoscopy in the Queen Mary Hospital are invited to participate in this prospective randomized study. Patients are excluded if they are unable to provide informed consent or have undergone previous colorectal resection, or have personal history of colorectal cancer, inflammatory bowel disease, familial adenomatous polyposis, Peutz-Jeghers syndrome, or other polyposis syndromes. Patients who are considered to be unsafe for polypectomy including patients with bleeding tendency and those with severe comorbid illnesses will be excluded. In addition, patients are excluded post-randomization if either the cecum could not be intubated for various reasons or Boston Bowel Preparation Scale (BBPS) score is <2.

Study design and randomization:

This is a prospective randomized crossover trial comparing the proximal adenoma detection rate and miss rate of BLI (ELUXEO endoscopic system) vs NBI (290 video system) vs WLI which is conducted in the Endoscopy Center of the Queen Mary Hospital of Hong Kong. Eligible patients are randomly allocated to four groups in a 1:1:1 ratio to undergo tandem colonoscopy of the proximal colon, defined as cecum to splenic flexure. The three groups are: (1) NBI follow by WLI; (2) BLI follow up WLI; (3) WLI follow by WLI. Randomization will be carried out by computer generated random sequences and stratified according to endoscopist's experiences (experienced versus fellows) and indications of colonoscopy (symptomatic vs screening/surveillance). All procedures are performed with high-definition endoscopes. The patients are blinded to the group assignment.

ELIGIBILITY:
Inclusion Criteria:

* Age 40 or above
* scheduled for colonoscopy

Exclusion Criteria:

* unable to provide informed consent
* have undergone previous colorectal resection,
* personal history of colorectal cancer, inflammatory bowel disease, familial adenomatous polyposis, Peutz-Jeghers syndrome, or other polyposis syndromes.
* Patients who are considered to be unsafe for polypectomy including patients with bleeding tendency and those with severe comorbid illnesses
* poor bowel preparation

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 884 (Actual)
Dates: Start 2018-11-08 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Proximal adenoma detection rate | one day
  proportion of patients with proximal adenoma detected on first examination

SECONDARY OUTCOMES:
proximal polyp detection rate | one day
  proportion of patients with proximal polyp detected on first examination
proximal adenoma miss rate | one day
  proportion of patients with proximal adenoma detected on second examination
proximal polyp miss rate | one day
  proportion of patients with proximal polyp detected on second examination

CONTACTS AND LOCATIONS:
Overall Officials: Wai Keung Leung, MD, Principal Investigator — The University of Hong Kong
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Leung WK, Tsui VWM, Mak LL, Cheung MK, Hui CK, Lam CP, Wong SY, Liu KS, Ko MK, To EW, Guo CG, Lui TK. Blue-light imaging or narrow-band imaging for proximal colonic lesions: a prospective randomized tandem colonoscopy study. Gastrointest Endosc. 2023 Nov;98(5):813-821.e3. doi: 10.1016/j.gie.2023.06.004. Epub 2023 Jun 10. PMID 37307902